CLINICAL TRIAL: NCT07250243
Title: Turkish Validity and Reliability Study of the John Hopkins In-Room Independence Scale: A Cross-Sectional Diagnostic Value Study
Brief Title: Turkish Validation and Reliability of the John Hopkins In-Room Independence Scale
Status: Enrolling by invitation | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, MD, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 08.19.2025/approval no: 5022
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Independence; Hemiplegia; Paraplegia; Parkinson Disease; Polyneuropathy; Arthrosis; Amputation; Musculoskeletal Disease
Keywords: independence; in-room independence; musculoskeletal disease
MeSH Terms: conditions — Hemiplegia; Paraplegia; Parkinson Disease; Polyneuropathies; Osteoarthritis; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving treatment in a physical medicine and rehabilitation inpatient clinic: Patients aged 18 and over who are receiving inpatient treatment at the PM&R inpatient clinic with any diagnosis
  Interventions: Other: In-room independence assessment

INTERVENTIONS:
Other: In-room independence assessment — The Turkish validity and reliability study of The Johns Hopkins Hospital In-Room Independence Scale(JH-IRIS) will be conducted.The researchers who developed the scale were contacted and a two-stage translation was conducted based on their suggestions.The final Turkish version of the scale was agreed upon after an online meeting with the developing research group.Because the other scales used in the original study lacked Turkish validity, the decision was made to use the Turkish-validated Morse and Henrich-2 Fall Scales and the Barthel Index, with the research team's permission.The study planned to include patients hospitalized for rehabilitation over a four-month period, regardless of their indication.This will allow comparison with previously validated Turkish fall risk and independence scales.One week later, patients will complete the JH-IRIS again and undergo a test-retest.The scale will be evaluated by two different researchers to determine inter-observer reliability.

SUMMARY:
The aim was to conduct a Turkish validity and reliability study of the Johns Hopkins In-Room Independence Scale. We believe this scale will address the lack of information regarding fall risk and dependency, particularly for patients scheduled for discharge and their caregivers.

DETAILED DESCRIPTION:
Independence and fall risk are critical for many illnesses and age groups. Patients receiving inpatient physical therapy in a Physical Medicine and Rehabilitation clinic often worry about returning home and performing daily activities after discharge. Therefore, this scale assessing in-room independence will allow us to better warn and guide patients about potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over
* Volunteering to participate in the study

Exclusion Criteria:

* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and over who are receiving inpatient treatment in the PM&R service with any diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Johns Hopkins Hospital In-Room Independence Scale | 1 week
  The Johns Hopkins Hospital In-Room Independence Scale is a scale that assesses a person's in-room independence, assessing mobility, toileting, and cognition. It consists of 15 items. A person who passes all items receives a score of 15. Failure on any item indicates in-room dependency.

SECONDARY OUTCOMES:
Morse Fall Scale | 1 week
  The Morse Fall Scale is an 125-point assessment tool that evaluates the risk of falling by considering factors such as fall history, secondary diagnoses, need for a walking aid, gait and transfer, and mental status; higher scores indicate poorer functioning.
Hendrich II Fall Risk Scale | 1 week
  The Hendrich II Fall Risk Scale assesses patients' fall risk. The scale includes factors like confusion, depression, dizziness, male gender, certain medications, and a mobility test. A score of 5 or above indicates high risk.
Barthel Index | 1 week
  The Barthel Index is an evaluation tool used to measure independence in performing 10 physical activities of daily living, with a primary focus on self-care and mobility. Minimum: 0,. Maximum: 100 (higher is better).

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Study Chair — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided